CLINICAL TRIAL: NCT04705675
Title: The Impact of Breastfeeding Education on Breastfeeding Behavior and the Use of Traditional Practices (An Example From Turkey): A Randomized Controlled Trial
Brief Title: The Impact of Breastfeeding Education on Breastfeeding Behavior and the Use of Traditional Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Durmaz (Other)
Responsible Party: Sponsor-Investigator, Aysegul Durmaz, Asst. Prof., Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Breas. Trad. Pra.
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Breastfeeding; Breasfeeding Traditional Practices; Post Procedural Discharge
Keywords: Breastfeeding; Education; Behavior; Traditional practices
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Intervention Model Description: The study was designed to be parallel group, randomized controlled study (1:1). Power was calculated using the GPower 3.1 program. In the power analysis performed at a confidence interval of 95% and a margin of error of plus/minus 5%, sample size was calculated as a total of 304 mothers with 152 in the study group and 152 in the control group.A total of 304 mothers were evenly and homogeneously assigned to both groups.
Who Masked: Participant
Masking Description: Participants didn't know which group they were allocated. The participants will be blind when they attend breastfeeding education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The mothers in the experimental group (152) were administered.
  Interventions: Behavioral: Breastfeeding Education
- Control Group (No Intervention): The mothers in the control group (152) were administered.

INTERVENTIONS:
Behavioral: Breastfeeding Education — The mothers were asked to remember the pseudonyms they used on the pretest and to use the same pseudonym on the posttest. Following the pretest, the mothers in the study group were taken into a separate room at the FHC and asked to breastfeed their infants. The mothers' breastfeeding behaviors were observed. After the breastfeeding, each mother was provided an average 30-minute session of individual education. All of the mothers in the study group received the education from the same researcher. Both audio and visual materials were used in the mothers' training.
  Arms: Experimental Group

SUMMARY:
H1a: The breastfeeding education has an effect the behaviors of mothers toward breastfeeding.

H1b: The breastfeeding education has an effect on the use of traditional breastfeeding practices.

H0a: The breastfeeding education has not an effect the behaviors of mothers toward breastfeeding.

H0b: The breastfeeding education has not an effect on the use of traditional breastfeeding practices.

DETAILED DESCRIPTION:
The study was designed to be parallel group, randomized controlled study (1:1). The study universe consisted of all of the mothers presenting at the family health centers (FHC's) of a province in Turkey over the period February 1, 2018-October 31, 2018.

The study samples were included 152 study and 152 control group which individuals selected by simple random sampling.In the power analysis performed at a confidence interval of 95% and a margin of error of plus/minus 5%, sample size was calculated as a total of 304 mothers with 152 in the study group and 152 in the control group.

The researchers collected the data for the study. They administered the pretest and filled out the personal information form prior to the planned individual education. The mothers were asked to remember the pseudonyms they used on the pretest and to use the same pseudonym on the posttest. Following the pretest, the mothers in the study group were taken into a separate room at the FHC and asked to breastfeed their infants. The mothers' breastfeeding behaviors were observed. After the breastfeeding, each mother was provided an average 30-minute session of individual education. All of the mothers in the study group received the education from the same researcher. Both audio and visual materials were used in the mothers' training. The researchers educated the mothers on breastfeeding techniques in an effort to encourage them to develop the skill of correctly using the positions taught and then the mothers were asked to practice what they had learned. The researcher took care to be positive and support whenever the mother attempted the right move in breastfeeding while also providing encouraging feedback when something went wrong. Included in the content of the education were the topics of the formation of breast milk and its benefits, the duration of breastfeeding, the sufficiency of breast milk, factors that reduced and increased it, things to look out for before breastfeeding, taking the right position for breastfeeding and positioning the baby on the breast, the steps in breastfeeding, burping the baby afterwards, milking and storing the mother's milk, and other issues that could pose problems during breastfeeding (Turkish Ministry of Health Basic Health Services General Directorate 2008). To test the retention of what was learned in the training, a posttest was administered to the groups one month following the education.

The Personal Information Form and the Breastfeeding Behaviors and Traditional Practices Assessment Form were used as data collection tools.

Statistical analyses were performed using IBM SPSS (Statistical Package for Social Sciences) Statistics 22 software. Descriptive statistics (means, standard deviation, frequencies and percentages) were used in the analysis of the findings. Normality tests (Kolmogorov-Smirnov Test) were performed on all continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* To receive breasfeeding education
* To have singleton birth or one infant
* Not have complications postpartum period
* Not have chronic diseases or mental disorders
* Older than 18 years
* To voluntary to participate
* To know how to read, write and speak in Turkish
* To stay within this study until the end
* To have a newborn with no complications
* To have a 0-6 months healthy infants

Exclusion Criteria:

* Not receive breasfeeding education
* Having multiple birth or more than a baby
* Having complications postpartum period
* Having chronic diseases or mental disorders
* Younger than 18 years
* To refuse to participate
* Not knowing how to read, write and speak Turkish
* To leave early this study
* Having a newborn with complications
* Having a baby in need of medical care
* To have a older than 0-6 months infants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Pre-Education Mothers' traditional breastfeeding practices | 20 minute after the admittance to the family health centers
  The Breastfeeding Behaviors Form was created in line with the literature. The questionnaires were filled out by the researchers using the face-to-face interview method. The questionnaire for Breastfeeding Behaviors included the following questions: Education about mother's milk and breastfeeding, When did you first breastfeed your baby after birth? Have you given your baby the first milk from your breast? Has your baby been given any food other than breast milk after birth? Why are you giving other food to your baby? Have you continued to feed your baby any other food? Do you give your baby water after breastfeeding? Breastfeeding Length (Daily)-Frequency (Daily)-Position-Latching, Having Problems with Breastfeeding, b. How long do you intend to breastfeed your baby?
Pre-Education Breastfeeding behavior | 20 minute after the admittance to the family health centers
  Traditional Practices Assessment Form was created in line with the literature. The questionnaires were filled out by the researchers using the face-to-face interview method. The Mother's Traditional Breastfeeding Practices Assessment Form included the following questions: Are there any traditional practices you use for breastfeeding? Do you think the traditional Practices you use for breastfeeding are useful? Who suggested traditional practices regarding breastfeeding? Do you voluntarily use traditional breastfeeding practices? Are There Foods You Consume to Increase Breast Milk? Who recommended the foods you consume to increase breast milk? Do you think the Food You Consume to Increase Breast Milk is beneficial? Do you voluntarily consume the foods you consume to increase breast milk?

SECONDARY OUTCOMES:
Post-Education | 1 month following the breastfeeding education.
  The Breastfeeding Behaviors Form was created in line with the literature. The questionnaires were filled out by the researchers using the face-to-face interview method. The questionnaire for Breastfeeding Behaviors included the following questions: How are you feeding your baby now? Has your baby been given any food other than breast milk after birth? Breastfeeding Length (Daily)-Frequency (Daily)-Position-Latching, Having Problems with Breastfeeding, What do you pay attention to avoid cracked nipples in your breast? Why are you giving other food to your baby? Do you give your baby water after breastfeeding? How long do you intend to breastfeed your baby? Does your partner support your breastfeeding?
Post-Education | 1 month following the breasfeeding education.
  Traditional Practices Assessment Form was created in line with the literature. The questionnaires were filled out by the researchers using the face-to-face interview method. The Mother's Traditional Breastfeeding Practices Assessment Form included the following questions: Are there any traditional practices you use for breastfeeding? Do you think the traditional Practices you use for breastfeeding are useful? Who suggested traditional practices regarding breastfeeding? Do you voluntarily use traditional breastfeeding practices? Are There Foods You Consume to Increase Breast Milk? Who recommended the foods you consume to increase breast milk? Do you think the Food You Consume to Increase Breast Milk is beneficial? Do you voluntarily consume the foods you consume to increase breast milk?

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If study' IPD are used, my article should be cited.

REFERENCES:
- [Background] Zielinska MA, Sobczak A, Hamulka J. Breastfeeding knowledge and exclusive breastfeeding of infants in first six months of life. Rocz Panstw Zakl Hig. 2017;68(1):51-59. PMID 28303701
- [Background] Bellu R, Condo M. Breastfeeding promotion: evidence and problems. Pediatr Med Chir. 2017 Jun 28;39(2):156. doi: 10.4081/pmc.2017.156. PMID 28673077
- [Background] Huang P, Yao J, Liu X, Luo B. Individualized intervention to improve rates of exclusive breastfeeding: A randomised controlled trial. Medicine (Baltimore). 2019 Nov;98(47):e17822. doi: 10.1097/MD.0000000000017822. PMID 31764775
- [Background] Sharma A. Efficacy of early skin-to-skin contact on the rate of exclusive breastfeeding in term neonates: a randomized controlled trial. Afr Health Sci. 2016 Sep;16(3):790-797. doi: 10.4314/ahs.v16i3.20. PMID 27917213
- [Background] Sandoval Jurado L, Jimenez Baez MV, Olivares Juarez S, de la Cruz Olvera T. [Breastfeeding, complementary feeding and risk of childhood obesity]. Aten Primaria. 2016 Nov;48(9):572-578. doi: 10.1016/j.aprim.2015.10.004. Epub 2016 Feb 12. Spanish. PMID 26880166
- [Background] McFadden A, Gavine A, Renfrew MJ, Wade A, Buchanan P, Taylor JL, Veitch E, Rennie AM, Crowther SA, Neiman S, MacGillivray S. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2017 Feb 28;2(2):CD001141. doi: 10.1002/14651858.CD001141.pub5. PMID 28244064
- [Background] Hay G, Baerug AB. The benefits of exclusive breastfeeding up to six months. Tidsskr Nor Laegeforen. 2019 May 3;139(9). doi: 10.4045/tidsskr.19.0105. Print 2019 May 28. No abstract available. English, Norwegian. PMID 31140258
- [Background] Del Ciampo LA, Del Ciampo IRL. Breastfeeding and the Benefits of Lactation for Women's Health. Rev Bras Ginecol Obstet. 2018 Jun;40(6):354-359. doi: 10.1055/s-0038-1657766. Epub 2018 Jul 6. PMID 29980160